CLINICAL TRIAL: NCT00976209
Title: A Randomized, Two-Way Crossover, Multicenter, Consumer Preference Study of Two Oral Formulations of Phenylephrine Hydrochloride.
Brief Title: Consumer Preference Study of Two Formulations of Phenylephrine Hydrochloride (Study CL2008-15)(P07530)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 18122; CL2008-15; P07530 (Other: Merck)
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2011-03-25 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Vasomotor Rhinitis; Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Vasomotor; Rhinitis, Allergic, Seasonal | interventions — Phenylephrine; Tablets; Oxymetazoline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenylephrine Hydrochloride Extended Release Tablets, 30 mg (Experimental)
  Interventions: Drug: Phenylephrine Hydrochloride (HCl) Extended Release (ER) Tablets 30 mg
- Phenylephrine Hydrochloride Immediate Release Tablets, 10 mg (Active Comparator)
  Interventions: Drug: Phenylephrine Hydrochloride (HCl) Immediate Release (IR) tablets, 10 mg

INTERVENTIONS:
Drug: Phenylephrine Hydrochloride (HCl) Extended Release (ER) Tablets 30 mg — Phenylephrine HCl ER tablets 30 mg taken every 12 hours, twice daily, for 3 days.
  Arms: Phenylephrine Hydrochloride Extended Release Tablets, 30 mg
Drug: Phenylephrine Hydrochloride (HCl) Immediate Release (IR) tablets, 10 mg — Phenylephrine HCl IR tablets 10 mg taken every four hours (no more than 6 times daily) for 3 days.
  Other Names: Sudafed PE®
  Arms: Phenylephrine Hydrochloride Immediate Release Tablets, 10 mg

SUMMARY:
This is a randomized, two-way crossover, multicenter study evaluating the consumer preference of Phenylephrine Extended Release Tablets, 30 mg to be taken as one tablet every 12 hours, or Phenylephrine Immediate Release Tablets, 10 mg to be taken as one tablet every 4 hours in subjects with at least mild allergic rhinitis and nasal congestion. Approximately 250 participants will complete a questionnaire after taking one test product for 3 days followed by a 3 day (± 1 day) washout period; and then taking the alternate test product for 3 days. Analysis of which product the consumer preferred, if any, and which product was more convenient, if any, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers must be 18 years or older.
* Participants must be willing to stop use of current decongestant and allergy medications during the study, and at the start of the run-in period (Visit 2).
* Participants must have a documented history of allergic rhinitis caused by ragweed allergen for at least the prior two years.
* Participants must have a documented skin testing (prick with wheal >= 3 mm larger than the diluent or intradermal with wheal >=7 mm larger than the diluent control) or a positive in vitro test for specific IgE to the ragweed allergen within the last four years.
* Participants must have signs by clinical evaluation and symptoms of nasal congestion of at least mild severity (sign/symptom clearly present, but minimal awareness; easily tolerated) at Visit 3 following the run-in period and at visit 5 following the washout period.
* Clinical laboratory tests (complete hematology, blood chemistries, urinalysis) must be within normal limits or clinically acceptable to the Investigator/Sponsor. Sponsor will not grant waivers.
* Participants must have a seated (after 5 minutes of rest) systolic/diastolic blood pressure ≤ 138/88 mmHg.
* Participants must have normal or clinically acceptable physical exam and electrocardiogram (ECG) on 12-lead ECG (recorded at 25 mm/s).
* Participants must be free of any clinically significant disease that requires a physician's care and/or would interfere with study evaluations, procedures or participation.
* Participants must agree not to take monoamine oxidase inhibitor (MAOI) for 14 days before study participation and 14 days after the end of the study.
* Participants must be willing to give written informed consent (prior to any study related procedures being performed) and able to adhere to restrictions and examination schedules.
* Female participants of childbearing potential (a non-menopausal female who has not had a hysterectomy, bilateral oophorectomy, or medically documented ovarian failure, including a young woman who has not yet started menstruating) must be using medically acceptable (documented failure rate of less than 1%) birth control measures. Examples of medically acceptable contraception include hormonal contraceptives, intrauterine device (IUD), double-barrier method (any combination of male or female condom, diaphragm, spermicidal gel, sponge) or sterilization.
* Participants must be able to read and write English, and must understand the dosing schedule.

Exclusion Criteria:

* Participants must not have any significant medical condition which, in the judgment of the investigator, is a contraindication to the use of phenylephrine HCl, might interfere with the study or requires treatment expected to affect the blood pressure. These may include thyroid disease (e.g. hyperthyroidism, hypothyroidism), uncontrolled diabetes mellitus, coronary heart disease, ischemic heart disease, elevated intraocular pressure, prostatic hypertrophy, etc.
* Participants that have received allergen immunotherapy or Xolair (omalizumab) therapy within the past two years.
* Participants who have a history of any clinically significant local or systemic infectious disease within four weeks prior to initial treatment administration.
* Participants who have participated in a clinical trial of an investigational treatment within 30 days prior to the start of the study (Run-in Period Day 1).
* Participants who are, appear to be, or are known to be, current or former addicts or alcoholics.
* Participants who have a known allergy or intolerance to phenylephrine HCl, any other decongestant, loratadine, desloratadine or any other antihistamine.
* Females who are pregnant, nursing or unwilling to use/practice medically acceptable contraception (documented failure rate of less than 1%).
* Participants with a history of asthma, rhinitis medicamentosa, or acute or chronic sinusitis.
* Participants that have used use of inhaled, oral, rectal, topical, intramuscular, and/or intravenous potent chronic or intermittent corticosteroids (up to 1% topical hydrocortisone is permitted).
* Participants who work at the study site and/or for the Investigator or are family members of study staff and/or the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenylephrine HCl 30 ER First, Then Phenylephrine HCl 10 IR: Participants received a 5-day run in period with Loratadine 10 mg tablets until the end of the second treatment period. Participants received Phenylephrine Hydrochloride (HCl) 30 mg Extended Release (ER) tablets every 12 hours, twice daily, for 3 days. After a 3 day (+/- 1 day) washout period, participants were crossed over and received Phenylephrine HCl 10 mg Immediate Release (IR) tablets, every 4 hours (no more than 6 times daily) for 3 days.
- Phenylephrine HCl 10 IR First, Then Phenylephrine HCl 30 ER: Participants received a 5-day run in period with Loratadine 10 mg tablets until the end of the second treatment period. Participants received Phenylephrine Hydrochloride 10 mg Immediate Release tablets, every 4 hours (no more than 6 times daily) for 3 days. After a 3 day (+/- 1 day) washout period, participants were crossed over and received Phenylephrine Hydrochloride 30 mg Extended Release tablets every 12 hours, twice daily, for 3 days.
Period: Treatment Period 1
Arm/Group | Phenylephrine HCl 30 ER First, Then Phenylephrine HCl 10 IR | Phenylephrine HCl 10 IR First, Then Phenylephrine HCl 30 ER
Started | 165 | 166
Completed | 162 | 165
Not Completed | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other | 0 | 1
Period: Wash-out Period
Arm/Group | Phenylephrine HCl 30 ER First, Then Phenylephrine HCl 10 IR | Phenylephrine HCl 10 IR First, Then Phenylephrine HCl 30 ER
Started | 162 | 165
Completed | 158 | 163
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 1 | 0
Period: Treatment Period 2
Arm/Group | Phenylephrine HCl 30 ER First, Then Phenylephrine HCl 10 IR | Phenylephrine HCl 10 IR First, Then Phenylephrine HCl 30 ER
Started | 158 | 163
Completed | 158 | 161
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenylephrine HCl 30 ER First, Then Phenylephrine HCl 10 IR | Phenylephrine HCl 10 IR First, Then Phenylephrine HCl 30 ER | Total
Number analyzed (Participants) | 165 | 166 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (11.07) | 38.3 (11.45) | 39.5 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 103 | 214
  Male | 54 | 63 | 117

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Preferred Phenylephrine HCl 30 mg Extended Release Tablets, as Compared to Phenylephrine HCl 10 mg Immediate Release Tablets for the Relief of Nasal Congestion
Description: Preference was calculated based on total participants that completed the study.
  Responses to the following questions in the consumer preference questionnaire were the basis for the preference endpoints:
  Which product, if any, did you prefer for the relief of nasal congestion?
  The possible answers were:
  * I preferred the relief of Treatment A (the every 12 hours white tablet; Phenylephrine HCl 30 mg Extended Release Tablet)
  * I preferred the relief of Treatment B (the every 4 hours red tablet; Phenylephrine HCl 10 mg Immediate Release tablet)
  or
  • I did not have a preference
Time Frame: Visit 6 (Period 2, Day 4)
Population: A total of 319 of 331 subjects who completed both treatment periods provided a response to the primary endpoint, and hence were included in the Modified Intent-to-Treat (MITT) population.
Measure: Number; unit: Percentage of participants
Groups:
- All Participants: Participants received Phenylephrine HCl ER tablets 30 mg taken every 12 hours, twice daily, for 3 days and Phenylephrine HCl IR tablets 10 mg taken every four hours (no more than 6 times daily) for 3 days in a cross-over fashion. A 3 day (+/- 1 day) washout period separated the two treatment periods.
Arm/Group | All Participants
Number analyzed (Participants) | 319
Percentage of participants
  Phenylephrine HCL ER, 30 mg | 55
  Phenylephrine HCl IR, 10 mg | 28
  No Preference | 17

2. Secondary Outcome: Percentage of Participants That Preferred the Convenience of Phenylephrine HCl 30 mg Extended Release Tablets, as Compared to Phenylephrine HCl 10 mg Immediate Release Tablets
Description: Convenience was calculated based on total participants that completed the study.
  Responses to the following questions in the consumer preference questionnaire were the basis for the preference endpoints:
  Secondary Endpoint
  Which product, if any, was more convenient?
  The possible answers were:
  * I preferred the convenience of Treatment A (the every 12 hours white tablet; Phenylephrine HCl 30 mg Extended Release Tablet)
  * I preferred the convenience of Treatment B (the every 4 hours red tablet; Phenylephrine HCl 10 mg Immediate Release tablet)
  or
  • I did not have a preference
Time Frame: Visit 6 (Period 2, Day 4)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 319
Percentage of participants
  Phenylephrine HCL ER, 30 mg | 88
  Phenylephrine HCL IR, 10 mg | 6
  No Preference | 6

ADVERSE EVENTS:
Description: Participants who had taken at least one dose of treatment were included in the safety population. 7 participants discontinued (d/c) prior to receiving Phenylephrine IR 10 mg and were not included. 3 participants d/c prior to receiving Phenylephrine HCl ER 30 mg and 1 additional participant returned all medication without use and were not included.
Groups:
- Phenylephrine HCl ER, 30 mg: Phenylephrine Hydrochloride (HCl) Extended Release (ER) tablets 30 mg taken every 12 hours, twice daily, for 3 days.
- Phenylephrine HCl IR, 10 mg: Phenylephrine Hydrochloride (HCl) Immediate Release tablets 10 mg taken every four hours (no more than 6 times daily) for 3 days.
Arm/Group | Phenylephrine HCl ER, 30 mg | Phenylephrine HCl IR, 10 mg
Serious Adverse Events (participants affected / at risk) | 0/327 | 0/324
Other Adverse Events (participants affected / at risk) | 0/327 | 0/324

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No